CLINICAL TRIAL: NCT00003665
Title: Phase I Trial of a Dendritic Cell Vaccine for Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02292; UPCC-4697; NCI-T98-0033; CDR0000066759 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

ARMS (3):
- Arm I (Experimental): Patients receive 3 different doses of peptide pulsed DC vaccine IV, each divided into 3 different peptide pulsed pools administered over 30 minutes.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine; Biological: gp100 antigen; Biological: therapeutic tumor infiltrating lymphocytes; Biological: tyrosinase peptide
- Arm II (Experimental): Patients receive 3 different doses of peptide pulsed DC vaccine subcutaneously/intradermally to sites with no evidence of disease. At the lowest dose, patients receive 3 different peptide pulsed pools, each administered at a separate site. At the higher doses, patients receive 3 injections further subdivided into 6 and administered at 6 distinct sites.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine; Biological: gp100 antigen; Biological: therapeutic tumor infiltrating lymphocytes; Biological: tyrosinase peptide
- Arm III (Experimental): Patients receive peptide pulsed DC vaccine intranodally in groin or ancillary lymph nodes at the lower 2 doses of the 3 administered to arms I and II. At the lower dose, patients receive 3 different peptide pulsed pools, each administered into a different node. At the higher dose, patients receive 3 injections further subdivided into 6 and administered at 6 distinct sites.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine; Biological: gp100 antigen; Biological: therapeutic tumor infiltrating lymphocytes; Biological: tyrosinase peptide

INTERVENTIONS:
Biological: dendritic cell-MART-1 peptide vaccine
Biological: gp100 antigen
Biological: therapeutic tumor infiltrating lymphocytes
Biological: tyrosinase peptide

SUMMARY:
Randomized phase I trial to study the effectiveness of vaccine therapy in treating patients who have stage IV melanoma. Vaccines may make the body build an immune response to kill tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the dose-limiting toxicities, maximum tolerated dose, recommended phase II dose, and rate of sensitization of T cells at each dose level in patients with melanoma receiving dendritic cell vaccine.

II. Determine the overall (complete and partial) response rate, duration of response, and optimal route of administration in this patient population.

OUTLINE: This is a dose escalation study. Patients are randomized to one of three treatment arms.

All patients undergo leukopheresis to obtain lymphocyte and myeloid origin mononuclear cell fractions for preparation of dendritic cell (DC) vaccine. In each arm, cohorts of up to 5 patients receive escalating doses of vaccine. The maximum tolerated dose (MTD) is defined as the dose preceding that at which 2 or more of 5 patients experience dose-limiting toxicity. Randomization ceases if the MTD has been reached in 2 arms, although accrual may continue. Treatment repeats every 2 weeks for a total of 4 doses.

Arm I: Patients receive 3 different doses of peptide pulsed DC vaccine IV, each divided into 3 different peptide pulsed pools administered over 30 minutes.

Arm II: Patients receive 3 different doses of peptide pulsed DC vaccine subcutaneously/intradermally to sites with no evidence of disease. At the lowest dose, patients receive 3 different peptide pulsed pools, each administered at a separate site. At the higher doses, patients receive 3 injections further subdivided into 6 and administered at 6 distinct sites.

Arm III: Patients receive peptide pulsed DC vaccine intranodally in groin or ancillary lymph nodes at the lower 2 doses of the 3 administered to arms I and II. At the lower dose, patients receive 3 different peptide pulsed pools, each administered into a different node. At the higher dose, patients receive 3 injections further subdivided into 6 and administered at 6 distinct sites.

Patients are followed at 2 weeks and then monthly for 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

-Histologically confirmed stage IV melanoma Must be MHC Class I HLA-A2.1

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-1
* Life expectancy: At least 2 months
* Platelet count at least 100,000/mm3
* INR no greater than 1.5 mg/dL
* No coagulopathies including thrombocytopenia
* Partial thromboplastin time no greater than 50 seconds
* No major cardiac illness
* No major respiratory illness
* No active systemic infection or other illness
* No peripheral vascular disease
* Not pregnant or nursing
* Effective contraception required of all fertile patients during and for one month after completion of treatment

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior immunotherapy
* No concurrent immunotherapy
* At least 30 days since prior chemotherapy
* No concurrent chemotherapy
* At least 30 days since prior radiotherapy
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1999-04; Primary Completion 2002-10 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Czerniecki, MD, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania, United States